CLINICAL TRIAL: NCT01771471
Title: A Phase II, Randomized, Double Blind, Placebo Controlled Study Evaluating the Treatment of Degenerative Lumbar Discs With Allogeneic Cultured Chondrocytes
Brief Title: A Study Comparing the Safety and Effectiveness of Cartilage Cell Injected Into the Lumbar Disc as Compared to a Placebo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in clinical strategy
Sponsor: ISTO Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISTO-NUQ02-10-12-00
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2016-09

CONDITIONS: Degenerative Disc Disease
Keywords: back pain; intervertebral disc; lumbar spine
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NuQu treatment (Experimental): single administration
  Interventions: Biological: NuQu
- Saline (Other): single administration
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NuQu — Allogenic juvenile chondrocytes (NuQu) in fibrin carrier.
  Arms: NuQu treatment
Other: Placebo — 0.9% w/v Sodium Chloride for Injection, USP
  Arms: Saline

SUMMARY:
This is a clinical study to collect safety and preliminary efficiency information on the use of NuQu chondrocytes (cartilage cells) delivered to the center of a lumbar spinal disc to treat low back pain.

DETAILED DESCRIPTION:
This is a Phase II clinical study to collect additional safety data and preliminary efficiency of juvenile chondrocytes, delivered in fibrin carrier (NuQu®) to the nucleus of lumbar intervertebral discs for the treatment of discogenic pain. This to be accomplished through a double blinded, placebo-controlled study of clinically meaningful endpoints including validated, subject reported outcomes of pain and disability, health related quality of life and subject satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent and must sign the Institutional Review Board approved Informed Consent Form;
* Is at least 21 years of age;
* Have central low back pain aggravated by movement and or postural changes (standing/sitting);
* Have had back pain for at least 6 months, and have failed conservative management
* One Grade III or IV (Pfirrmann Scale) degenerated lumbar disc;

Exclusion Criteria:

* Current disc extrusion at any level in their lumbar spine; disc bulges or protrusions at any level in the lumbar spine resulting in nerve root compression;
* Severe disc narrowing (equal to or more than 50% loss of disc height at the targeted level);
* Type II or III Modic changes at any level;
* Type I Modic changes at any level other than the targeted level;
* Type I Modic changes at the treated level if maximum height of the changes is 25% or more of the vertebral body height;
* Osteoporotic compression fracture at any vertebral level;
* Lumbar Scheurmann's disease;
* Antero or retrolisthesis ≥ 3mm at any level;
* Currently experiencing chronic pain generating from any other source, which (in the judgment of the investigator) may interfere with the evaluation of back pain, and or disability;
* Infection at the planned treatment site, history of systemic or local infection, which (in the investigator's judgment) may compromise subject participation and/or safety;
* Currently diagnosed with immune-deficiency, which in the investigator's opinion may compromise subject participation and/or safety;
* Receiving any immune-suppressant therapies other than short term steroid preparations;
* BMI≥40;
* Diagnosed with any comorbid conditions including: abnormal bleeding, AIDS, diabetes, hepatic or renal disease, and cardiopulmonary disorders such as COPD, MI and CHF; active malignancy or history of malignancy, or diseases of bone metabolism, which in the investigator's opinion may compromise subject participation and/or safety;
* Has a history of alcoholism, medication or intravenous drug abuse, psychosis, is a prisoner, has a personality disorder(s), poor motivation, emotional or intellectual issues that would likely make the subject unreliable for the study, or 3 or more Waddell Signs of nonorganic Behavior or any combination of variables in the Investigator's judgment that should exclude a potential subject;
* Has pending litigation against a health care professional, except where required by the insurer as a condition of coverage, personal injury compensation or litigation claims;
* Has active or pending workers' compensation claims;
* Has contraindications for MRI.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-11; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | 12 months

SECONDARY OUTCOMES:
Subject Satisfaction as measured by subject's willingness to have the same procedure for the same condition | 24 Months
  Success to be measured by the response of "Definitely True" or "Mostly True" to the following: "All things considered I would have the treatment again for the same condition".
MRI | 24 Months
Visual Analog Scale | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Domagoj Coric, MD, Principal Investigator — Carolina Neurosurgery and Spine Associates
Locations (10):
- United States (10):
  - Alabama Orthopedic and Spine Center, Birmingham, Alabama
  - California Spine Diagnostics, San Francisco, California
  - The Spine Institute, Center for Spinal Restoration, Santa Monica, California
  - Ortho Georgia, Macon, Georgia
  - Tufts University School of Medicine, Newton, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - The NeuroSpine Institute, Eugene, Oregon
  - Spine Team Texas, Southlake, Texas
  - Spinal Reseach Foundation, Reston, Virginia